CLINICAL TRIAL: NCT06114927
Title: Validation of the Spanish Version of the Conceptualization of Pain Questionnaire
Acronym: COPAQ-S
Status: Completed | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Principal Investigator, University Rovira i Virgili
Other Study IDs: Ceim: 114/2018
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Child Development; Pain; Adolescent Behavior
Keywords: survey; children; health knowledge; chronic pain; pain education
MeSH Terms: conditions — Pain; Adolescent Behavior; Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: To answer a 15-question survey.
  Interventions: Behavioral: Validation of a questionnaire

INTERVENTIONS:
Behavioral: Validation of a questionnaire — The Conceptualization of Pain Questionnaire (COPAQ-S) Spanish version consist of 15 items and asks respondents to respond if they believe the items/statements to be true or false, although they are allowed to respond undecided. A score of 0 is given to incorrect responses and those marked as undecided; the sum of all the correct answers gives the total score. The higher the score, the better the participant understands the concept of pain.

SUMMARY:
The goal of this observational study is to develop a questionnaire to assess a child's concept of pain and to evaluate its psychometric properties in schoolchildren aged 8-17 years. The main question[s] it aims to answer are:

* Validate to Spanish language the Conceptualization of Pain Questionnaire to assess a child's concept of pain.
* Conduct an analysis to evaluate its psychometric properties. Participants will respond a questionnaire of 15 items and asks respondents to respond if they believe the items/statements to be true or false, although they are allowed to respond undecided.

DETAILED DESCRIPTION:
The inclusion criteria were: to be able to read and write in Spanish language and excluded if they suffered from an intellectual disability that, according to the teachers, could interfere with their participation in the study procedures.

The main outcome was: The Conceptualization of Pain Questionnaire - Spanish version.

ELIGIBILITY:
Inclusion Criteria:

* Were able to read and write in Spanish

Exclusion Criteria:

* If they suffered from an intellectual disability that, according to the teachers, could interfere with their participation in the study procedures.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Schoolchildren aged 8-17 years.
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The Conceptualization of Pain Questionnaire (COPAQ-S) Spanish version. | 1 year
  It consist of 15 items and asks respondents to respond if they believe the items/statements to be true or false, although they are allowed to respond undecided. A score of 0 is given to incorrect responses and those marked as undecided; the sum of all the correct answers gives the total score. The higher the score, the better the participant understands the concept of pain.

SECONDARY OUTCOMES:
Age | 1 year
  Years
Gender | 1 year
  Female, male
School Year | 1 year
  Years

CONTACTS AND LOCATIONS:
Locations (1):
- Rovira i Virgili University, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No